CLINICAL TRIAL: NCT01313221
Title: A Randomized, Blinded Assessor Study to Evaluate the Efficacy and Safety of Etanercept 50 mg Once Weekly Plus As Needed Topical Agent Versus Etanercept 50 mg Twice Weekly in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: Efficacy and Safety of Etanercept 50 mg Once Weekly Plus As Needed Topical Agent in Moderate to Severe Plaque Psoriasis
Acronym: REFINE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20090647
Record Dates: First submitted 2011-02-24; First posted 2011-03-11 (Estimated); Results first posted 2014-05-02 (Estimated); Last update posted 2017-03-15 (Actual); Status verified 2017-02

CONDITIONS: Psoriasis
Keywords: plaque psoriasis; moderate; severe; etanercept; Enbrel; topical
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular | interventions — Etanercept; Anti-Infective Agents, Local

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- Etanercept 50 mg BIW (Active Comparator): Following 12 weeks of etanercept 50 mg twice weekly, participants were randomized to 50 mg etanercept twice weekly for 12 weeks.
  Interventions: Biological: etanercept
- Etanercept 50 mg QW + Topical (Experimental): Following 12 weeks of etanercept 50 mg twice weekly, participants were randomized to 50 mg etanercept once weekly plus as needed topical agents.
  Interventions: Biological: etanercept; Drug: Topical agents

INTERVENTIONS:
Biological: etanercept — Administered by subcutaneous injection
  Other Names: Enbrel
Drug: Topical agents — Topical agents prescribed at the discretion of the Principal Investigator and were are limited to the following:
  * hydrocortisone 2.5%
  * betamethasone valerate 0.1%
  * betamethasone dipropionate 0.05%
  * clobetasol 0.05%
  * calcitriol
  * calcipotriol plus betamethsone dipropionate 0.05%
  Arms: Etanercept 50 mg QW + Topical

SUMMARY:
To estimate the difference in effectiveness between treatment with etanercept 50 mg twice weekly (BIW) and treatment with etanercept 50 mg once weekly (QW) plus an as needed (PRN) topical agent for 12 weeks in adults with moderate to severe plaque psoriasis.

DETAILED DESCRIPTION:
The recommended starting dose of etanercept for adult plaque psoriasis patients is a 50 mg dose given twice a week (BIW) for 3 months followed by a reduction to a maintenance dose of 50 mg once weekly (QW). While most patients with moderate to severe plaque psoriasis are managed satisfactorily on etanercept monotherapy, a proportion may require a modified or alternative treatment regimen (eg, to handle flares or loss of effect) at some point during their chronic management. Despite the clinical need, no published data from randomized controlled studies are currently available that demonstrate efficacy and safety of combined etanercept-based regimens in patients with plaque psoriasis.

The addition of an as-needed topical medication to the step-down dose of etanercept 50 mg once weekly administered after the initial 12 week period of 50 mg twice weekly may be a potential option for patients who may require adjunctive therapy. This study aimed to provide data on this treatment option by estimating the difference in mean percent change in Psoriasis Area and Severity Index (PASI) scores between step-down etanercept 50 mg once weekly supplemented with as-needed topical medication and continuous treatment with etanercept 50 mg twice weekly.

Eligible patients will be enrolled in the study and will receive etanercept 50 mg twice weekly for 12 weeks. After 12 weeks of etanercept treatment, participants will be randomized in a 1:1 ratio to 1 of 2 treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Has had stable moderate to severe plaque psoriasis for at least 6 months (eg, no morphology changes or significant flares of disease activity in the opinion of the investigator).
* Has a body surface area (BSA) involvement ≥ 10% and Psoriasis Area and Severity Index (PASI) ≥ 10 at screening and at baseline.
* Is a candidate for systemic therapy or phototherapy in the opinion of the investigator.
* Other inclusion criteria may apply.

Exclusion Criteria:

* Has active guttate, erythrodermic, or pustular psoriasis at the time of the screening visit.
* Has evidence of skin conditions at the time of the screening visit (eg, eczema) that would interfere with evaluations of the effect of etanercept on psoriasis.
* Diagnosed with medication-induced or medication-exacerbated psoriasis.
* Significant concurrent medical conditions.
* Has any active localized infection; requiring local intervention or chronic or localized infections.
* Other exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2011-04; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (20):
- Canada (20):
  - Research Site, Calgary, Alberta
  - Research Site, Surrey, British Columbia
  - Research Site, Vancouver, British Columbia
  - Research Site, Winnipeg, Manitoba
  - Research Site, Moncton, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Courtice, Ontario
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Markham, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, North Bay, Ontario
  - Research Site, Peterborough, Ontario
  - Research Site, Richmond Hill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Waterloo, Ontario
  - Research Site, Windsor, Ontario
  - Research Site, Montreal, Quebec
  - Research Site, Québec, Quebec
  - Research Site, Saint-Hyacinthe, Quebec

REFERENCES:
- [Background] Papp KA, Barber K, Bissonnette R, Bourcier M, Lynde CW, Poulin Y, Shelton J, Garces K, Toole J, Poulin-Costello M. Improvements in patient-reported outcomes in patients with psoriasis receiving etanercept plus topical therapies: results from REFINE. J Eur Acad Dermatol Venereol. 2015 Aug;29(8):1555-61. doi: 10.1111/jdv.12934. Epub 2015 Jan 21. PMID 25611084
- [Background] Papp KA, Barber K, Bissonnette R, Bourcier M, Lynde CW, Poulin Y, Shelton J, Toole J, Vieira A, Poulin-Costello M. A Randomized, blinded assessor study to Evaluate the efFIcacy and safety of etanercept 50 mg once weekly plus as Needed topical agent vs. Etanercept 50 mg twice weekly in patients with moderate to severe plaque psoriasis (REFINE). J Eur Acad Dermatol Venereol. 2015 Feb;29(2):361-366. doi: 10.1111/jdv.12555. Epub 2014 Jul 1. PMID 24980988
- [Background] Gooderham MJ, Poulin-Costello M, Shelton J, Bayan N, Papp KA. Predictors of Topical Use in Psoriasis Patients in the REFINE Study. J Cutan Med Surg. 2016 Mar-Apr;20(2):106-12. doi: 10.1177/1203475415604322. Epub 2015 Sep 1. PMID 26330052
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrollment :29 April 2011; last patient enrollment: 4 June 2012.
Pre-assignment Details: A total of 414 patients were screened,310 patients were enrolled and 287 randomized in this study; 144 in the etanercept monotherapy group (group A) and 143 in the etanercept plus an as-needed topical agent group (group B). 23 patients were not randomized because they did not complete the 12-week open-label treatment period before randomization.
Groups:
- Etanercept 50 mg BIW: Following 12 weeks of etanercept 50 mg twice weekly (BIW), participants were randomized to 50 mg etanercept by subcutaneous injection twice weekly for 12 weeks.
- Etanercept 50 mg QW + Topical: Following 12 weeks of etanercept 50 mg twice weekly, participants were randomized to 50 mg subcutaneous injection once weekly (QW) plus as needed topical agents.
- Non-randomized: Enrolled participants received etanercept 50 mg twice weekly but discontinued prior to completing the 12-week open-label treatment period.
Period: Overall Study
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical | Non-randomized
Started | 144 | 143 | 23
Randomized | 144 | 143 | 0
Completed | 132 | 135 | 0
Not Completed | 12 | 8 | 23
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Non-compliance | 3 | 0 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 5
Not completed — Requirement for alternative therapy | 0 | 1 | 1
Not completed — Lost to Follow-up | 6 | 3 | 1
Not completed — Other | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 7
Not completed — Disease progression | 0 | 0 | 2
Not completed — Physician Decision | 0 | 0 | 2
Not completed — Pregnancy | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical | Non-randomized | Total
Number analyzed (Participants) | 144 | 143 | 23 | 310
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.7 (13.1) | 46.3 (14.6) | 36.6 (11.2) | 45.3 (13.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 46 | 49 | 14 | 109
  Male | 98 | 94 | 9 | 201
Race/Ethnicity, Customized [Number; unit: participants]
  American Indian or Alaska Native | 1 | 0 | 0 | 1
  Asian | 14 | 5 | 0 | 19
  Mixed Race | 1 | 0 | 0 | 1
  White | 120 | 130 | 22 | 272
  Other | 8 | 8 | 1 | 17
Body Mass Index (BMI) [Number; unit: participants]
  ≤ 30 | 81 | 80 | 13 | 174
  > 30 | 63 | 63 | 10 | 136
Prior anti-Tumor Necrosis Factor (TNF) Treatment [Number; unit: participants] — Based on participants in the Efficacy Evaluable set, all randomized participants, who had taken at least 1 dose of study drug and had at least 1 postrandomization efficacy evaluation (140 and 142 particiapants in each randomized treatment group respectively).
  participants
    Prior exposure | 24 | 22 | NA — Not reported for non-randomized participants | NA — Total not calculated because data are not available (NA) in one or more arms.
    Naive | 116 | 120 | NA — Not reported for non-randomized participants | NA — Total not calculated because data are not available (NA) in one or more arms.

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Psoriasis Area and Severity Index (PASI) From Week 12 to Week 24
Description: The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Change from Week 12 to Week 24 is presented as a percentage of the Week 12 value: Week 12 value - Week 24 value / Week 12 value * 100 so that a positive change indicates improvement. Change was adjusted for treatment using a mixed model.
Time Frame: Week 12 and Week 24
Population: Efficacy Evaluable set, which included all randomized participants who had taken at least 1 dose of study drug and had at least 1 post-randomization efficacy evaluation, and with available data at Week 12 and Week 24.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 139 | 140
percent change | 17.02 (7.06) | 0.86 (7.06)
Statistical Analysis 1: Comparison: Etanercept 50 mg BIW vs Etanercept 50 mg QW + Topical; Test type: Superiority or Other; Mean Difference (Final Values) = 16.16, 95% CI 2-sided [-3.50 to 35.82], Standard Error of Mean 9.99 — Adjusted for treatment in a mixed model

2. Secondary Outcome: Percent Change in PASI From Week 12 to Weeks 16 and 20
Description: The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Change from Week 12 presented as a percentage of the Week 12 value: Week 12 value - postbaseline value / Week 12 value * 100, so that a positive change indicates improvement. Change was adjusted for treatment using a mixed model.
Time Frame: Week 12, Week 16 and Week 20
Population: Efficacy Evaluable set with available data at each time point (indicated by n)
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 140 | 142
percent change
  Change from Week 12 to Week 16 (n=136, 137) | 16.03 (5.89) | 4.80 (5.87)
  Change from Week 12 to Week 20 (n=139, 140) | 19.79 (6.74) | 3.23 (6.74)
Statistical Analysis 1: Comparison: Etanercept 50 mg BIW vs Etanercept 50 mg QW + Topical; Difference in change from Week 12 to Week 16; Test type: Superiority or Other; Mean Difference (Final Values) = 11.23, 95% CI 2-sided [-5.13 to 27.60], Standard Error of Mean 8.31
Statistical Analysis 2: Comparison: Etanercept 50 mg BIW vs Etanercept 50 mg QW + Topical; Difference in change from Week 12 to Week 20; Test type: Superiority or Other; Mean Difference (Final Values) = 16.56, 95% CI 2-sided [-2.21 to 35.32], Standard Error of Mean 9.53

3. Secondary Outcome: Percent Change in PASI From Baseline to Weeks 12, 16, 20, and 24
Description: The Psoriasis Area and Severity Index (PASI) score is a combination of the intensity of psoriasis, assessed by the erythema (reddening), induration (plaque thickness) and desquamation (scaling) on a scale from none (0), mild (1), moderate (2), severe (3) or very severe (4), together with the percentage of the area affected, rated on a scale from 0 to 6. PASI scoring is performed at four body areas, the head, arms, trunk, and legs. The total PASI score ranges from 0 to 72. The higher the total score, the more severe the disease. Change from Baseline is presented as a percentage of the Baseline value: Baseline value - postbaseline value / Baseline value * 100, so that a positive change indicates improvement.
Time Frame: Baseline and Weeks 12, 16, 20, and 24
Population: Full analysis set, (all enrolled participants who had taken at least 1 dose of study treatment and had at least 1 post-baseline efficacy evaluation) and with available data. Last Observation Carried Forward (LOCF) imputation was used.
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
percent change
  Change at Week 12 (n=143, 142) | 62.12 (28.62) | 65.48 (28.59)
  Change at Week 16 (n=138, 138) | 68.25 (27.08) | 72.67 (25.06)
  Change at Week 20 (n=142, 141) | 70.98 (27.43) | 73.25 (25.35)
  Change at Week 24 (n=142, 141) | 71.71 (27.56) | 72.56 (27.76)

4. Secondary Outcome: Percentage of Participants With a PASI 50 Response
Description: The percentage of participants with a 50% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI score is based on an assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and the percent area affected as observed on the day of examination. The score ranges from 0 (best outcome) to 72 (worst outcome).
Time Frame: Baseline and Weeks 12, 16, 20 and 24
Population: Full analysis set with a non-missing response; LOCF was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
percentage of participants
  Week 12 (n=143, 142) | 71.3 [63.9 to 78.7] | 75.4 [68.3 to 82.4]
  Week 16 (n=138, 138) | 76.1 [69.0 to 83.2] | 86.2 [80.5 to 92.0]
  Week 20 (n=142,141) | 80.3 [73.7 to 86.8] | 86.5 [80.9 to 92.2]
  Week 24 (n=142, 141) | 78.2 [71.4 to 85.0] | 88.7 [83.4 to 93.9]

5. Secondary Outcome: Percentage of Participants With a PASI 75 Response
Description: The percentage of participants with a 75% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI score is based on an assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and the percent area affected as observed on the day of examination. The score ranges from 0 (best outcome) to 72 (worst outcome).
Time Frame: Baseline and Weeks 12, 16, 20 and 24
Population: Full analysis set with a non-missing response; LOCF was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
percentage of participants
  Week 12 (n=143, 142) | 44.1 [35.9 to 52.2] | 52.1 [43.9 to 60.3]
  Week 16 (n=138, 138) | 52.2 [43.8 to 60.5] | 58.7 [50.5 to 66.9]
  Week 20 (n=142,141) | 54.9 [46.7 to 63.1] | 58.9 [50.7 to 67.0]
  Week 24 (n=142, 141) | 59.2 [51.1 to 67.2] | 60.3 [52.2 to 68.4]

6. Secondary Outcome: Percentage of Participants With a PASI 90 Response
Description: The percentage of participants with a 90% reduction (improvement) in Psoriasis Area and Severity Index (PASI) score from Baseline. PASI score is based on an assessment of erythema (reddening), induration (plaque thickness), desquamation (scaling), and the percent area affected as observed on the day of examination. The score ranges from 0 (best outcome) to 72 (worst outcome).
Time Frame: Baseline and Weeks 12, 16, 20 and 24
Population: Full analysis set with a non-missing response; LOCF was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
percentage of participants
  Week 12 (n=143, 142) | 17.5 [11.3 to 23.7] | 12.7 [7.2 to 18.1]
  Week 16 (n=138, 138) | 23.2 [16.1 to 30.2] | 22.5 [15.5 to 29.4]
  Week 20 (n=142,141) | 28.9 [21.4 to 36.3] | 22.0 [15.1 to 28.8]
  Week 24 (n=142, 141) | 32.4 [24.7 to 40.1] | 27.0 [19.6 to 34.3]

7. Secondary Outcome: Percentage of Participants With a Static Physician's Global Assessment (sPGA) of Psoriasis Score of 0 (Clear) or 1 (Almost Clear)
Description: The sPGA scale is completed by the same blinded assessor performing the PASI assessments and is designed to evaluate the physician's global assessment of the participant's psoriasis based on severity of induration, scaling, and erythema. The sPGA is assessed on a scale of 0 to 5 (0 = clear, 5 = severe).
Time Frame: Weeks 12, 16, 20, and 24
Population: Full Analysis Set, LOCF was used.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
percentage of participants
  Week 12 (n=143, 142) | 40.6 [32.5 to 48.6] | 45.8 [37.6 to 54.0]
  Week 16 (n=139, 139) | 50.4 [42.0 to 58.7] | 50.4 [42.0 to 58.7]
  Week 20 (n=142, 141) | 51.4 [43.2 to 59.6] | 48.9 [40.7 to 57.2]
  Week 24 (n=142, 141) | 53.5 [45.3 to 61.7] | 45.4 [37.2 to 53.6]

8. Secondary Outcome: Percent Change in the Percentage of Body Surface Area (BSA) Involvement From Week 12 to Weeks 16, 20, and 24
Description: The percentage of body surface area involved with psoriasis was measured by the same blinded assessor performing the PASI assessments. Change from Week 12 is presented as a percentage of the Week 12 value: Week 12 value - postbaseline value / Week 12 value * 100, so that a positive change indicates improvement.
  Change was adjusted for treatment using a mixed model.
Time Frame: Weeks 12, 16, 20, and 24
Population: Efficacy analysis set with available data
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 140 | 142
percent change
  Change from Week 12 to Week 16 (n=135, 138) | 18.77 (5.77) | 12.83 (5.72)
  Change from Week 12 to Week 20 (n=138, 140) | 22.89 (7.65) | 16.04 (7.61)
  Change from Week 12 to Week 24 (n=138, 140) | 15.60 (10.17) | 10.71 (10.15)

9. Secondary Outcome: Percent Change in the Percentage of Body Surface Area (BSA) Involvement From Baseline to Weeks 12, 16, 20, and 24
Description: The percentage of body surface area involved with psoriasis was measured by the same blinded assessor performing the PASI assessments.
  Change from Baseline \ is presented as a percentage of the Baseline value: Baseline value - postbaseline value / Baseline value * 100, so that a positive change indicates improvement.
Time Frame: Baseline and Weeks 12, 16, 20, and 24
Population: Full analysis set with available data; LOCF was used
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
percent change
  Change at Week 12 (n=142, 142) | 58.13 (33.18) | 62.47 (36.10)
  Change at Week 16 (n=138, 139) | 65.75 (30.95) | 72.88 (27.90)
  Change at Week 20 (n=142, 141) | 70.37 (30.30) | 75.86 (26.70)
  Change at Week 24 (n=142, 141) | 71.80 (29.72) | 75.39 (29.52)

10. Secondary Outcome: Change From Week 12 to Week 24 in Dermatology Quality of Life Index (DQLI) Total Score
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. Change from Week 12 to Week 24 is calculated as: Week 12 value - Week 24 value so that a positive change indicates improvement. Change was adjusted for treatment using a mixed model.
Time Frame: Week 12 and Week 24
Population: Efficacy Evaluable set with available data
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 134 | 127
units on a scale | 0.52 (0.38) | -0.03 (0.39)

11. Secondary Outcome: Change From Baseline to Weeks 12 and 24 in Dermatology Quality of Life Index (DQLI) Total Score
Description: The DLQI questionnaire asks participants to evaluate the degree that psoriasis has affected their quality of life in the last week, and includes the following parameters: symptoms and feelings, daily activities, leisure activities, work or school activities, personal relationships and treatment related feelings. Participants answer 10 questions on a scale from 0 (not at all) to 3 (very much); the range of the total score is 0 to 30. A score of 21 to 30 means an extremely large effect on the participant's life whereas 0-1 means that the disease has no effect at all. Change from Baseline was calculated as Baseline value - postbaseline value so that a positive change indicates improvement.
Time Frame: Baseline and Week 12 and Week 24
Population: Full analysis set with available data; LOCF was used
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
units on a scale
  Change at Week 12 (n=141, 139) | 10.01 (7.03) | 9.71 (6.15)
  Change at Week 24 (n=135, 129) | 10.71 (7.80) | 9.87 (6.91)

12. Secondary Outcome: Change in Treatment Satisfaction Questionnaire for Medications (TSQM) Scores From Week 12 to Week 24
Description: TSQM is a validated questionnaire consisting of 14 questions regarding a participant's perception of the level of satisfaction or dissatisfaction with the medication they are taking. Four scales are generated: side effects, effectiveness, convenience, and global satisfaction. Optional responses are: Extremely Dissatisfied, Very Dissatisfied, Dissatisfied, Somewhat Satisfied, Satisfied, Very Satisfied, and Extremely Satisfied. From the responses, a scale score from 0 - 100 is calculated, with a higher score indicating greater satisfaction. Change was calculated as Week 24 - Week 12 so that a positive change indicates improvement over time. Change was adjusted for treatment using a mixed model.
Time Frame: Week 12 and Week 24
Population: Efficacy Evaluable with available data; n indicates the number of patients with available data for each scale.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 140 | 142
units on a scale
  Effectiveness (n=135, 127) | -3.05 (2.64) | 0.09 (2.74)
  Convenience (n=135, 128) | -1.27 (1.19) | 2.57 (1.23)
  Side effects (n=135, 126) | -0.43 (1.30) | 2.22 (1.35)
  Global Satisfaction (n=135, 128) | -4.09 (1.59) | 1.34 (1.64)

13. Secondary Outcome: Change in Treatment Satisfaction Questionnaire for Medications (TSQM) Scores From Baseline to Weeks 12 and 24
Description: The TSQM is a validated questionnaire consisting of 14 questions regarding a participant's perception of the level of satisfaction or dissatisfaction with the medication they are taking. Four scales are generated: side effects, effectiveness, convenience, and global satisfaction. Optional responses are: Extremely Dissatisfied, Very Dissatisfied, Dissatisfied, Somewhat Satisfied, Satisfied, Very Satisfied, and Extremely Satisfied. From the responses, a scale score from 0 - 100 is calculated, with a higher score indicating greater satisfaction. Change was calculated as postbaseline value - Baseline value so that a positive change indicates improvement.
Time Frame: Baseline and Weeks 12 and 24
Population: Full analysis set; LOCF was used; n indicates the number of patients with available data for each scale at each time point.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
units on a scale
  Week 12: Effectiveness (n=133, 129) | 31.37 (34.50) | 32.64 (36.66)
  Week 12: Convenience (n=132, 129) | 15.87 (26.86) | 16.47 (30.39)
  Week 12: Side effects (n=132, 125) | 0.0 (19.07) | -0.15 (20.75)
  Week 12: Global Satisfaction (n=133, 129) | 31.10 (32.99) | 27.09 (32.48)
  Week 24: Effectiveness (n=127, 120) | 27.08 (36.10) | 32.45 (40.29)
  Week 24: Convenience (n=127, 121) | 14.83 (25.88) | 18.53 (29.00)
  Week 24: Side effects (n=127, 119) | -0.74 (22.04) | 1.26 (19.44)
  Week 24: Global Satisfaction (n=128, 120) | 26.73 (32.54) | 28.39 (35.94)

14. Secondary Outcome: Health Resource Utilization: Number of Participants With Visits to a Healthcare Provider
Description: Participants completed a questionnaire to assess their health resource utilization (HRU) related to psoriasis. To assess the number of visits to a healthcare provider, participants answered the following questions regarding the past 4 weeks: How many times have you been to any physician's office or urgent care clinic? How many times have you seen a nurse practitioner, a physician assistant, a psychologist, a naturopath, an acupuncturist, a chiropractor, or other healthcare professional (HCP)? The number of participants with one or more visits is reported.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set with available data; LOCF was used.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline: Any Physician Visit (n=137, 135) | 52 | 45
  Week 24: Any Physician Visit (n=131, 124) | 28 | 25
  Baseline: Nurse Practitioner Visits (n=126, 130) | 9 | 14
  Week 24: Nurse Practitioner Visits (n=121, 116) | 3 | 9
  Baseline: Physician Assistant Visits (n=123, 124) | 10 | 8
  Week 24: Physician Assistant Visits (n=123, 113) | 7 | 5
  Baseline: Psychologist Visits (n=122, 125) | 1 | 2
  Week 24: Psychologist Visits (n=121, 112) | 1 | 2
  Baseline: Naturopath Visits (n=125, 125 | 4 | 2
  Week 24: Naturopath Visits (n=121, 111) | 1 | 2
  Baseline: Acupuncturist Visits (n=122, 125) | 0 | 1
  Week 24: Acupuncturist Visits (n=121, 111) | 2 | 2
  Baseline: Chiropractor Visits (n=124, 125) | 6 | 5
  Week 24: Chiropractor Visits (n=122, 112) | 7 | 9
  Baseline: Other HCP Visits (n=31, 42) | 12 | 20
  Week 24: Other HCP Visits (n=25, 35) | 6 | 11

15. Secondary Outcome: Health Resource Utilization: Number of Participants With Home Healthcare Visits
Description: Participants completed a questionnaire to assess their health resource utilization (HRU) related to psoriasis. To assess the number of homecare visits, participants answered the following question regarding the past 4 weeks: How many times have you received care from a health professional in your home? The number of participants with one or more visits is reported.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set with available data; LOCF was used.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline: Homecare Visits (n=138, 135) | 1 | 2
  Week 24: Homecare Visits (n=133, 127) | 1 | 1

16. Secondary Outcome: Health Resource Utilization: Number of Participants Requiring Paid Help With Chores
Description: Participants completed a questionnaire to assess their health resource utilization (HRU) related to psoriasis. To assess the number of participants who needed paid help with chores, participants answered the following question regarding the past 4 weeks: How many times have you paid someone to help you do chores around the house (cleaning, maintenance, lawn care)? The number of participants who paid for help one or more times is reported.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set with available data; LOCF was used.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline (n=134, 135) | 12 | 13
  Week 24 (n=132, 127) | 5 | 5

17. Secondary Outcome: Health Resource Utilization: Number of Participants Who Needed Friend or Family Care
Description: Participants completed a questionnaire to assess their health resource utilization (HRU) related to psoriasis. Participants answered the following question regarding the past 4 weeks: How many hours have you had a friend or family member take time off work to provide care or transportation? The number of participants who had paid or non-paid help for one or more hours is reported.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set with available data; LOCF was used.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline: Provided Paid Work (n=123, 121) | 5 | 6
  Week 24: Provided Paid Work (n=118, 113) | 7 | 6
  Baseline: Provided Non-paid Work (n=120, 124) | 6 | 8
  Week 24: Provided Non-paid Work (n=118, 114) | 4 | 4

18. Secondary Outcome: Health Resource Utilization: Out of Pocket Expenses
Description: Participants completed a questionnaire to assess their health resource utilization (HRU) related to psoriasis. To assess out of pocket expenses, participants answered the following question regarding the past 4 weeks: Not counting study mandated visits, what out-of-pocket expenses did you spend for the management of psoriasis (i.e. costs due to travelling to doctor appointment, hospital or clinic parking costs, alternative medications)?
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set with available data; LOCF was used.
Measure: Median (Inter-Quartile Range); unit: Canadian dollars
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
Canadian dollars
  Baseline (n=129, 132) | 1.0 [0.0 to 70.0] | 0.0 [0.0 to 50.0]
  Week 24 (n=117, 120) | 0.0 [0.0 to 3.0] | 0.0 [0.0 to 3.1]

19. Secondary Outcome: Health Resource Utilization: Employment Status
Description: Participants completed a questionnaire to assess their health resource utilization (HRU) related to psoriasis. Participants were asked their employment status at Baseline and at Week 24.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set; LOCF was used.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline: Employed full time | 81 | 72
  Baseline: Employed part time | 26 | 21
  Baseline: Unemployed | 16 | 21
  Baseline: Retired | 19 | 28
  Baseline: Unknown/Missing | 2 | 1
  Week 24: Employed full time | 81 | 67
  Week 24: Employed part time | 21 | 19
  Week 24: Unemployed | 16 | 13
  Week 24: Retired | 18 | 30
  Week 24: Unknown/Missing | 8 | 14

20. Secondary Outcome: Health Resource Utilization: Productivity While Working
Description: Participants who were employed were asked: How much did your psoriasis affect your productivity while you were working? Possible responses were: a) A great deal; b) Quite a bit; c) Somewhat; d) Minimally; e) Not at all.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set who were employed and with available data at each time point; LOCF was used. For the Etanercept 50 mg BIW group there were 106 and 100 participants with available data at Baseline and Week 24 respectively. For the Etanercept + Topical group there were 93 and 85 participants respectively.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline: A great deal | 7 | 6
  Baseline: Quite a bit | 16 | 13
  Baseline: Somewhat | 37 | 28
  Baseline: Minimally | 20 | 21
  Baseline: Not at all | 26 | 25
  Week 24: A great deal | 1 | 3
  Week 24: Quite a bit | 4 | 1
  Week 24: Somewhat | 7 | 12
  Week 24: Minimally | 24 | 12
  Week 24: Not at all | 64 | 57

21. Secondary Outcome: Health Resource Utilization: Number of Participants With Missed Hours From Work
Description: Participants who were employed answered the following question regarding the past 4 weeks: How many hours per week did you miss from work because of your psoriasis? The number of participants with one or more missed hours of work per week is reported.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set who were employed and with available data; LOCF was used.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline: Hours Missed From Work (n=101, 92) | 15 | 19
  Week 24: Hours Missed From Work (n=96, 83) | 5 | 6

22. Secondary Outcome: Health Resource Utilization: Ability to Perform Daily Activities
Description: Participants were asked: How much did your psoriasis affect your ability to do your daily activities or household chores? Possible answers were: a) A great deal; b) Quite a bit; c) Somewhat; d) Minimally; e) Not at all.
Time Frame: Baseline and 24 weeks
Population: Full Analysis Set; LOCF was used.
Measure: Number; unit: participants
Arm/Group | Etanercept 50 mg BIW | Etanercept 50 mg QW + Topical
Number analyzed (Participants) | 144 | 143
participants
  Baseline: A great deal | 11 | 11
  Baseline: Quite a bit | 14 | 16
  Baseline: Somewhat | 23 | 27
  Baseline: Minimally | 29 | 25
  Baseline: Not at all | 34 | 30
  Baseline: Unknown/Missing | 33 | 34
  Week 24: A great deal | 2 | 2
  Week 24: Quite a bit | 5 | 6
  Week 24: Somewhat | 9 | 7
  Week 24: Minimally | 16 | 7
  Week 24: Not at all | 56 | 64
  Week 24: Unknown/Missing | 56 | 57

23. Secondary Outcome: Number of Participants With Adverse Events
Description: An adverse event (AE) is defined as any untoward medical occurrence in a clinical trial participant. A serious adverse event is defined as an adverse event that meets at least 1 of the following serious criteria: • fatal, • life threatening, • requires in-patient hospitalization or prolongation of existing hospitalization, • results in persistent or significant disability/incapacity, • congenital anomaly/birth defect, and/or • other significant medical hazard.
Time Frame: 32 weeks
Population: Safety analysis was based on treatment received, regardless of group assignment. 177 patients are included in group A, including 144 patients randomized to group A, 23 patients who were non-randomized and 10 patients randomized to group B but never received topical agents; Group B includes 133 patients who received etanercept plus ≥1 topical agent.
Measure: Number; unit: participants
Groups:
- Etanercept Monotherapy: All participants who received etanercept at any time during the study, who never used a topical agent, regardless of treatment assignment, including those participants who were not randomized at Week 12.
- Etanercept + Topical: All participants who used a topical agent at least once during the study, regardless of treatment group assignment.
Arm/Group | Etanercept Monotherapy | Etanercept + Topical
Number analyzed (Participants) | 177 | 133
participants
  Any adverse event | 112 | 92
  Serious adverse event | 4 | 0
  AE leading to discontinuation of study treatment | 11 | 0
  AE leading to discontinuation from study | 8 | 0
  Fatal adverse event | 0 | 0

ADVERSE EVENTS:
Time Frame: 32 weeks
Description: Safety analysis was based on treatment received, regardless of group assignment. 177 patients are included in group A, including 144 patients randomized to group A, 23 patients who were non-randomized and 10 patients randomized to group B but never received topical agents; Group B includes 133 patients who received etanercept plus ≥1 topical agent.
Arm/Group | Etanercept Monotherapy | Etanercept + Topical
Serious Adverse Events (participants affected / at risk) | 4/177 | 0/133
Other Adverse Events (participants affected / at risk) | 65/177 | 62/133
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept Monotherapy (N=177) | Etanercept + Topical (N=133)
Crohn's disease (Gastrointestinal disorders) | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0
Gastroenteritis (Infections and infestations) | 1 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Etanercept Monotherapy (N=177) | Etanercept + Topical (N=133)
Fatigue (General disorders) | 7 | 8
Injection site erythema (General disorders) | 13 | 7
Injection site haematoma (General disorders) | 2 | 7
Injection site reaction (General disorders) | 16 | 17
Nasopharyngitis (Infections and infestations) | 24 | 20
Upper respiratory tract infection (Infections and infestations) | 12 | 13
Headache (Nervous system disorders) | 19 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results aftercompletion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.